CLINICAL TRIAL: NCT03226470
Title: Safety Study of Transcription Activator-like Effector Nucleases T512 in HPV16-infected Subjects
Brief Title: Study of Targeted Therapy Using Transcription Activator-like Effector Nucleases in Cervical Precancerous Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Head of Cancer Biology center, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017TALEN-V02
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Human Papillomavirus-Related Malignant Neoplasm
Keywords: Transcription Activator-like Effector Nucleases; Human papillomavirus; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T512 group (Experimental): Subjects will receive suppository with T512 at 2 intervals for one month.
  Interventions: Biological: T512

INTERVENTIONS:
Biological: T512 — T512 suppository contain 500 µg of T512 and suppocire.
  Other Names: TALEN-T512

SUMMARY:
This is an single arm clinical study of the safety and efficacy of T512 to possibly treat cervical intraepithelial neoplasia(CIN).

DETAILED DESCRIPTION:
Persistent infection with high-risk human papillomavirus (HPVs),especially types 16 and 18,may lead to cervical intraepithelial neoplasia(CIN).HPVs expresses the oncoproteins E6 and E7, both of which play key roles in maintaining viral infection and promoting carcinogenesis. Previous studies showed that using designated TALENs (T27 and T512) targeted HPV16 E6 and E7 produced disruption of HPV16 E6 and E7 DNA, decreased the expression of E6 and E7 proteins, and induced cell apoptosis.

This study will evaluate the safety and efficacy of and T512 in treating HPV Persistency and HPV16-positive CIN.

ELIGIBILITY:
Inclusion Criteria:

* Documented HPV16 infection and integration.
* Married and fertile, no fertility requirements.
* The cervical transformation zone was type I or II, and the biopsy results under colposcopy suggested SIL.
* Without administration of hormone in the last six months
* Subjects must be meet the ethical requirements and have signed informed consent

Exclusion Criteria:

* Pregnancy and breast feeding
* Any bacterial vaginitis
* Any Fungal vaginitis
* Any sexually transmitted diseases
* Active drug or alcohol abuse
* Any HPV medications within the past 12 weeks
* Allergy to active or non active ingredients in the study of drugs
* Cardiac insufficiency
* Liver and renal insufficiency
* Hypertension and severe complications
* Serious illness in past 30 days
* Currently participating in another clinical trial or any prior gene therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Safety-Number of participants with Adverse Events | 6 months
  Number of participants who report adverse events as a measure of safety

SECONDARY OUTCOMES:
Change of HPV16 DNA titers | Baseline, 3 and 6 months
  Blood samples will be taken at the indicated times
Number of dysplastic cells mearsured by ThinPrep Pap Test | Baseline, 3 and 6 months
  From high-grade squamous intraepithelial lesion (HSIL) to Low-grade Squamous Intraepithelial Lesion (LSIL), or from LSIL to negative
Change of cervical histological results | Baseline and 6 months
  Colposcopy Biopsy will be conducted at the baseline and month 6 on each subject

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, M.D., Study Director — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Hu Z, Ding W, Zhu D, Yu L, Jiang X, Wang X, Zhang C, Wang L, Ji T, Liu D, He D, Xia X, Zhu T, Wei J, Wu P, Wang C, Xi L, Gao Q, Chen G, Liu R, Li K, Li S, Wang S, Zhou J, Ma D, Wang H. TALEN-mediated targeting of HPV oncogenes ameliorates HPV-related cervical malignancy. J Clin Invest. 2015 Jan;125(1):425-36. doi: 10.1172/JCI78206. Epub 2014 Dec 15. PMID 25500889